CLINICAL TRIAL: NCT00890747
Title: A Phase 1/Pharmacokinetic Study of Sunitinib in Patients With Cancer Who Also Have HIV and Are on HAART Therapy
Brief Title: Sunitinib Malate in Treating HIV-Positive Patients With Cancer Receiving Antiretroviral Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02208; NCI-2012-02208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-061 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-061 (Other: CTEP); U01CA121947 (NIH); NCT01727102 (obsolete NCT alias)
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2013-09

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Langerhans Cell Histiocytosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Aggressive NK-cell Leukemia; AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Malignancies; AIDS-related Small Noncleaved Cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Clear Cell Renal Cell Carcinoma; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; HIV Infection; HIV-associated Hodgkin Lymphoma; Intraocular Lymphoma; Isolated Plasmacytoma of Bone; Light Chain Deposition Disease; Mast Cell Leukemia; Myelodysplastic Syndrome With Isolated Del(5q); Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Myeloid/NK-cell Acute Leukemia; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Osteolytic Lesions of Multiple Myeloma; Peripheral T-cell Lymphoma; Plasma Cell Neoplasm; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Primary Systemic Amyloidosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Renal Cell Cancer; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Stage IV Renal Cell Cancer; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
Keywords: HIV Infections; treatment experienced
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Histiocytosis, Langerhans-Cell; Lymphoma, Extranodal NK-T-Cell; Leukemia, Large Granular Lymphocytic; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Carcinoma, Renal Cell; Thrombocythemia, Essential; HIV Infections; Intraocular Lymphoma; Leukemia, Mast-Cell; Chromosome 5q Deletion Syndrome; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Neoplasms, Plasma Cell; Polycythemia Vera; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of sunitinib malate in treating human immunodeficiency virus (HIV)-positive patients with cancer receiving antiretroviral therapy. Sunitinib malate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and to investigate the pharmacological interactions of administering sunitinib (sunitinib malate) in subjects with cancer who are also HIV positive on anti-retroviral regimens containing protease inhibitors and/or non-nucleoside reverse transcriptase inhibitors.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of sunitinib in treating non-acquired immunodeficiency syndrome (AIDS) defining cancers (NADCs) in these subjects.

II. To detect alterations in antiretroviral drug pharmacokinetics due to sunitinib.

III. To detect alterations in immune parameters, including total leukocyte count, cluster of differentiation (CD) 4 and viral load, during sunitinib therapy.

IV. To correlate variations in genes involved in sunitinib absorption, metabolism, and elimination, including cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), cytochrome P450, family 3, subfamily A, polypeptide 5 (CYP3A5), ATP-binding cassette, sub-family B (MDR/TAP), member 1 (ABCB1), and breast cancer resistance protein (ABCG2), with drug pharmacokinetics.

V. To explore the potential for pharmacological interactions between sunitinib and newer antiretroviral agents such as integrase and chemokine (C-C motif) receptor 5 (gene/pseudogene) (CCR5) inhibitors.

OUTLINE: This is a dose-escalation study.

Patients receive sunitinib malate orally (PO) daily on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven solid tumor or hematological malignancy, including:

  * Metastatic renal cell carcinoma
  * A solid tumor malignancy, including an NADC or an AIDS-defining malignancy, if the subject has progressed following standard therapy and/or other curative options are not available
  * A hematologic malignancy, except for blast-phase leukemia, for which effective standard therapy or other curative options are not available
* Serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme linked immunosorbent assay (ELISA), positive western blotting (Western Blot), or other federally approved licensed HIV test, or a detectable blood level of HIV ribonucleic acid (RNA), or a positive anti-HIV antibody test
* On stable anti-retroviral therapy for at least 4 weeks with a protease inhibitor (PI)-based or non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimen of at least three drugs, with no intention to change the regimen within 8 weeks after starting study drug

  * Patients who are on NNRTI and ritonavir PI-based therapy are eligible and will be enrolled in the ritonavir PI-based group (Group 3)
  * Patients who are on NNRTI and non-ritonavir PI-based therapy are eligible and will be enrolled in the non-ritonavir PI-based group (Group 2); NOTE: accrual to Group 2 will be closed upon approval of version 7.0 of the protocol
  * Patients who are on a highly active antiretroviral therapy (HAART) combination that includes neither a PI nor a NNRTI agent are eligible and will be enrolled in the NNRTI-based group (Group 1)
* CD4 count > 50 cells/uL
* Karnofsky performance status > 60%
* Women of child-bearing potential must have a negative pregnancy test within 7 days before initiation of study drug dosing; post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; male and female subjects of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug; (Note: a woman of childbearing potential is one who is biologically capable of becoming pregnant; this includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives)
* Hemoglobin >= 8.0 gm/dL
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Platelet count >= 100,000 /mm^3
* Creatinine within institutional normal limits or glomerular filtration rate (GFR) > 60 mL/min/m^2 (calculated by the Cockcroft-Gault equation), calculated as follows:

  * For males = (140 - age[years]) x (body weight [kg])/ (72) x (serum creatinine [mg/dL])
  * For females = 0.85 x male value
* Total bilirubin should be =< 1.5 times upper limit of normal (ULN); if, however, the elevated bilirubin is felt to be secondary to indinavir therapy, then subjects will be allowed on protocol if total bilirubin =< 3.5 mg/dL, provided that the direct bilirubin is =< 1.5 times ULN; if the elevated bilirubin is felt to be secondary to atazanavir therapy, then subjects will be allowed on protocol without any limit on the total bilirubin if the direct bilirubin is =< 1.5 times ULN
* Aspartate transaminase AST (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase ALT (serum glutamate pyruvate transaminase [SGPT]) < 2.5 times the ULN; unless subjects have liver metastases, in which case both AST and ALT must be =< 5 times ULN
* Life expectancy of 3 months or more
* Ability and willingness to give informed consent
* Subjects must in the opinion of the Investigator be capable of complying with this protocol

Exclusion Criteria:

* Concurrent active opportunistic infection (OI)
* Acute treatment for an infection or other serious medical illness within 14 days prior to study entry
* Receipt of antineoplastic therapy, including investigational drug or standard treatment, within 2 weeks of study entry; must be able to demonstrate adequate recovery from prior therapy-related toxicities
* Major surgery or radiation within 3 weeks prior to study entry
* Concurrent treatment with medications, other than antiretroviral drugs used to treat HIV infection, that are known to inhibit or induce CYP3A4
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Clinically significant cardiovascular disease, including uncontrolled hypertension (diastolic blood pressure >= 100 mmHg despite optimal medical therapy) or unstable angina
* A myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack, or pulmonary embolism within 6 months of study entry
* Abnormal left ventricular ejection fraction per institutional standards
* Ongoing ventricular cardiac dysrhythmias of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) grade >= 2
* Subjects with a history of serious ventricular arrhythmia (ventricular tachycardia [VT] or ventricular fibrillation [VF] >= 3 beats in a row)
* Serious cardiac arrhythmia requiring medication
* QTc interval > 500 msec
* Psychiatric illness that would limit compliance with study requirements
* Pre-existing thyroid abnormality that cannot be maintained with medication to keep measures of thyroid stimulating hormone within the normal range
* Female subjects who are pregnant or breast-feeding
* Another severe and/or life-threatening medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Grades 3, 4, and 5, treatment-related adverse events, graded according to the National Cancer Institute (NCI) CTCAE version 3.0 | Up to 30 days after completion of study treatment
  Results will be presented descriptively. Continuous data will be summarized for each cohort using descriptive statistics (N, mean, median, standard deviation, minimum, maximum, geometric mean, and % coefficient of variation [CV]).
Dose-limiting toxicity (DLT) defined as an adverse event that is possibly related to the study medication, graded according to the NCI CTCAE version 3.0 | 6 weeks
  Results will be presented descriptively. Continuous data will be summarized for each cohort using descriptive statistics (N, mean, median, standard deviation, minimum, maximum, geometric mean, and % coefficient of variation [CV]).

SECONDARY OUTCOMES:
Evaluation of response | Up to 30 days after completion of study treatment
  Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) (solid tumors), AIDS Clinical Trials Group (ACTG) (Kaposi's sarcoma [KS]), Cheson (lymphoma), Durie (multiple myeloma), or International Working Group for Response Criteria for acute leukemias criteria depending on the subject's primary disease.
Antiretroviral drug pharmacokinetics due to sunitinib malate | At baseline and at 1, 2, 3, 4, 5, 6, 7, 8, and 24 hours of days 1and 2
  Pharmacokinetic parameters within the individual groups will be compared using a Kruskall-Wallis test, Wilcoxon non-parametric test for paired data and Mann-Whitney test for unpaired data.
Alterations in immune parameters, including total leukocyte count, CD4, and viral load | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Deeken, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - AIDS - Associated Malignancies Clinical Trials Consortium, Rockville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University - Jewish, Saint Loius, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Result] Rudek MA, Moore PC, Mitsuyasu RT, Dezube BJ, Aboulafia D, Gerecitano J, Sullivan R, Cianfrocca ME, Henry DH, Ratner L, Haigentz M Jr, Dowlati A, Little RF, Ivy SP, Deeken JF. A phase 1/pharmacokinetic study of sunitinib in combination with highly active antiretroviral therapy in human immunodeficiency virus-positive patients with cancer: AIDS Malignancy Consortium trial AMC 061. Cancer. 2014 Apr 15;120(8):1194-202. doi: 10.1002/cncr.28554. Epub 2014 Jan 28. PMID 24474568
- [Derived] Rais R, Zhao M, He P, Xu L, Deeken JF, Rudek MA. Quantitation of unbound sunitinib and its metabolite N-desethyl sunitinib (SU12662) in human plasma by equilibrium dialysis and liquid chromatography-tandem mass spectrometry: application to a pharmacokinetic study. Biomed Chromatogr. 2012 Nov;26(11):1315-24. doi: 10.1002/bmc.2697. Epub 2012 Jan 18. PMID 22259028